CLINICAL TRIAL: NCT07158749
Title: Generalized and Domain-Specific Episodic Thinking for Smoking Cessation: An 8-Week Pilot and Feasibility Trial
Brief Title: Generalized and Domain-Specific Episodic Thinking for Smoking Cessation
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: Virginia Polytechnic Institute and State University (Other)
Collaborators: National Cancer Institute (NCI) (NIH); Roswell Park Comprehensive Cancer Center (Unknown)
Responsible Party: Principal Investigator, Jeffrey Stein, Assistant Professor, Virginia Polytechnic Institute and State University
Allocation: Randomized | Model: Factorial | Masking: Single | Purpose: Treatment
Other Study IDs: 24-1183; 1R21CA294049 (NIH)
Record Dates: First submitted 2025-08-20; First posted 2025-09-08 (Actual); Last update posted 2025-09-12 (Actual); Status verified 2025-09

CONDITIONS: Cigarette Smoking Behavior
Keywords: Cigarette smoking; episodic future thinking
MeSH Terms: conditions — Cigarette Smoking

STUDY DESIGN:
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (4):
- Generalized episodic future thinking (EFT) (Experimental): The Generalized EFT group will identify positive events that may occur at 6 future time points (1 month to 5 years). These may include a broad range of personally significant milestones (e.g., weddings, birthdays) or other events that participants are looking forward to (e.g., spending time with loved ones). Participants will also generate vivid text descriptions, or cues (transcribed in their own words), to prompt EFT in the natural environment. These cues, including emotional impacts, will be elicited using standardized questions: Who are you with? What are you doing? Where are you? How are you feeling?
  Participants will be prompted to engage in Generalized EFT in the natural environment.
  Interventions: Behavioral: Episodic Future Thinking (EFT); Behavioral: Generalized episodic thinking
- Domain-specific episodic future thinking (EFT) (Experimental): The Domain-Specific EFT group will complete an identical interview as the Generalized EFT group to identify positive future events, with one exception. Following initial cue generation, participants will be provided with descriptions of lung cancer symptoms (e.g., painful breathing; extreme fatigue; coughing up blood, phlegm, or mucus) and will be asked to visualize and include details related to this experience and their emotional impact in their revised cues. Thus, cancer-related symptoms occur in the context of otherwise positive, personally significant events to further highlight the impact of the diagnosis and to be consistent with Generalized EFT.
  Participants will be prompted to engage in Domain-Specific EFT in the natural environment.
  Interventions: Behavioral: Episodic Future Thinking (EFT); Behavioral: Domain-specific episodic thinking
- Generalized episodic recent thinking (ERT) (Placebo Comparator): The Generalized ERT interview will be identical to the one described for Generalized EFT, except participants will describe positive events they experienced in the last week.
  Participants will be prompted to engage in Generalized ERT in the natural environment.
  Interventions: Behavioral: Episodic Recent Thinking (ERT); Behavioral: Generalized episodic thinking
- Domain-specific episodic recent thinking (ERT) (Active Comparator): The Domain-Specific ERT interview will be identical to the one described for Domain-Specific EFT, except participants will describe positive events they experienced in the last week and will subsequently add detail as though they were experiencing symptoms of lung cancer.
  Participants will be prompted to engage in Domain-Specific ERT in the natural environment.
  Interventions: Behavioral: Episodic Recent Thinking (ERT); Behavioral: Domain-specific episodic thinking

INTERVENTIONS:
Behavioral: Episodic Future Thinking (EFT) — Participants will engage in EFT for 8 weeks, three times a day. Participants will receive three daily text messages. Each prompt will link to a custom web interface that guides participants to read and vividly imagine one of their cues, chosen randomly. Visit times and durations will be recorded.
  Arms: Domain-specific episodic future thinking (EFT); Generalized episodic future thinking (EFT)
Behavioral: Episodic Recent Thinking (ERT) — Participants will engage in ERT for 8 weeks, three times a day. Participants will receive three daily text messages. Each prompt will link to a custom web interface that guides participants to read and vividly imagine one of their cues, chosen randomly. Visit times and durations will be recorded.
  Arms: Domain-specific episodic recent thinking (ERT); Generalized episodic recent thinking (ERT)
Behavioral: Domain-specific episodic thinking — Content of the episodic thinking intervention will experiencing the symptoms of lung cancer during a broad range of personally meaningful, otherwise positive, events (e.g., social events, celebrations, spending times with friends and family).
  Arms: Domain-specific episodic future thinking (EFT); Domain-specific episodic recent thinking (ERT)
Behavioral: Generalized episodic thinking — Content of the episodic thinking intervention will include a broad range of personally meaningful, positive, events (e.g., social events, celebrations, spending times with friends and family).
  Arms: Generalized episodic future thinking (EFT); Generalized episodic recent thinking (ERT)

SUMMARY:
Cigarette smoking remains common, particularly in rural areas, despite ample evidence that smoking causes cancer and respiratory disease. Successful smoking cessation yields the majority of its health benefits (e.g., avoidance of lung cancer) after years of sustained behavioral change; however, people who smoke cigarettes tend to show elevated rates of delay discounting (i.e., devaluation of delayed outcomes) and a bias for immediate gratification. The overall goal of this project is to develop different versions of an episodic future thinking intervention (i.e., visualization of the future) and test their feasibility and efficacy for smoking cessation in rural and urban populations.

DETAILED DESCRIPTION:
Cigarette smoking causes more than a dozen cancers, including cancers of the head and neck, colon, bladder, and lung. Although quitting smoking drastically reduces the risk of cancer mortality, rates of cessation are low, particularly in rural areas and other communities. Current evidence-based treatments for smoking cessation have made progress, but substantial room for innovation remains and novel strategies are needed. Successful smoking cessation may be considered, in part, an intertemporal choice between continuing to smoke and achieving the delayed health benefits associated with quitting (e.g., avoidance of lung cancer). Thus, quitting requires one's behavior to be sufficiently motivated by future outcomes. Unfortunately, robust cross-sectional and longitudinal evidence indicates that people who smoke cigarettes show elevated delay discounting, or a bias for immediate gratification. Prior research shows that delay discounting predicts treatment failure and relapse in smoking cessation. These findings suggest that delay discounting often prevents successful quitting because the health benefits of cessation (e.g., avoiding cancer) are too delayed to motivate sustained behavioral change. Thus, delay discounting is a therapeutic target in smoking cessation, where interventions that increase valuation of future outcomes may facilitate quitting. Episodic future thinking (EFT) is one such scalable intervention that is designed to shift time perspective and reduce bias for immediate gratification by promoting vivid and frequent visualization of a broad range of personally significant future events (e.g., weddings, birthdays, spending time with loved ones). In laboratory studies, research has shown that this form of generalized EFT in cigarette smokers reduces delay discounting and motivation to smoke (i.e., cigarette consumption, craving, and valuation). Moreover, strong preliminary evidence suggests that cancer-related EFT, a novel form of the intervention that involves visualizing the future experience of smoking-related lung cancer, may be more efficacious for reducing urges to smoke than the generalized form. The proposed trial will adapt both forms of EFT (generalized and cancer-related) for clinical use in smoking cessation. Remote intervention delivery and outcomes assessment (breath carbon monoxide and number of cigarettes smoked per day) will be used to minimize clinical burden and increase intervention reach and access, including in rural populations who often lack access to evidence-based treatments for smoking cessation. In an eight-week proof-of-concept trial, participants will be prompted to engage in EFT or control episodic thinking multiple times per day and during acute craving episodes. Specific Aims 1 and 2 will examine the feasibility and efficacy, respectively, of generalized and cancer-related EFT to reduce smoking. An Exploratory Aim will investigate the potential moderating role of income, education, sex, and other characteristics (e.g., baseline delay discounting, cigarettes/day) in the effects of EFT on smoking outcomes.

ELIGIBILITY:
Inclusion Criteria:

* smoked cigarettes daily for the last 30 days;
* salivary cotinine > 30 ng/mL, consistent with tobacco use;
* plan to quit smoking in the next 30 days

Exclusion Criteria:

* prior diagnosis with a smoking-related illness (e.g., respiratory disease);
* past 30-day use any smoking cessation treatment;
* anxiety or mood disorders; and
* medical contraindications for use of nicotine replacement therapy (e.g. pregnancy).

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 134 (Estimated)
Dates: Start 2026-01-01 (Estimated); Primary Completion 2027-05-01 (Estimated); Study Completion 2027-05-01 (Estimated)

PRIMARY OUTCOMES:
Cigarettes smoked per day | From Week 0 to the end of treatment at 8 weeks
  A timeline followback questionnaire will be used to assess the number of cigarettes smoked per day. Lower values reflect better outcomes.

SECONDARY OUTCOMES:
Other tobacco/nicotine product use per day | From Week 0 to the end of treatment at 8 weeks
  A timeline followback questionnaire will be used to assess the number of times participants use other tobacco/nicotine products per day (excluding cigarettes and nicotine patch). Lower values reflect better outcomes.
7-day point prevalence cigarette abstinence | Week 8
  A timeline followback questionnaire will be used to assess cigarette abstinence status (binary) over the final seven days of the intervention.

OTHER OUTCOMES:
Nicotine patch adherence (feasibility outcome) | From Week 1 to the end of treatment at 8 weeks
  A timeline followback questionnaire will be used to assess frequency of use of the study-provided nicotine patches. Higher values reflect better adherence to nicotine replacement therapy.
Depressive symptoms (feasibility outcome) | From Week 0 to the end of treatment at 8 weeks
  Depression symptoms over the last 2 weeks will be assessed using the Patient Health Questionnaire-8 (PHQ-8). Total scores on this scale range from 0 (no depressive symptoms) to 24 (severe depressive symptoms).
Anxiety symptoms (feasibility outcome) | From Week 0 to the end of treatment at 8 weeks
  Anxiety symptoms over the last 2 weeks will be assessed using the Generalized Anxiety Disorder-7 (GAD-7) questionnaire. Total scores on this scale range from 0 (no anxiety symptoms) to 21 (severe anxiety symptoms).
Episodic thinking adherence (feasibility outcome) | From Week 1 to the end of treatment at 8 weeks
  Adherence to the episodic thinking interventions will be measured as the percentage of daily cue prompts that participants access.
Perceived convenience (feasibility outcome) | From Week 1 to the end of treatment at 8 weeks
  Participants will evaluate perceived convenience of the intervention, both overall and its individual components, using visual analog scales with ratings ranging from 0 to 100. Higher ratings reflect greater convenience
Perceived helpfulness (feasibility outcome) | From Week 1 to the end of treatment at 8 weeks
  Participants will evaluate perceived helpfulness of the intervention, both overall and its individual components, using visual analog scales with ratings ranging from 0 to 100. Higher ratings reflect greater helpfulness.

CONTACTS AND LOCATIONS:
Overall Officials: Jeffrey Stein, PhD, Principal Investigator — Virginia Polytechnic Institute and State University
Locations (1):
- Fralin Biomedical Research Institute at VTC, Roanoke, Virginia, United States

IPD SHARING:
Plan to Share IPD: Yes
All de-identified study data that are included in publication results will be shared using a project-specific url.
Supporting Information: SAP, ICF, Analytic Code
Time Frame: Study data and supporting information will be available beginning 3 months and ending 5 years after the publication of results.
Access Criteria: All shared deidentified study data and supporting information will be available without restriction via a project-specific url.